CLINICAL TRIAL: NCT04436406
Title: Measurement of PD-L1 Expression in Cancer to Monitor Treatment Response.
Brief Title: PD-L1 Expression in Cancer (PECan Study).
Acronym: PECan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: NanoMab Technology (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRAS 256684
Record Dates: First submitted 2020-03-09; First posted 2020-06-18 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Non-small Cell Lung Cancer; Melanoma
Keywords: immunotherapy; checkpoint inhibitors; molecular imaging; non-small cell lung cancer; melanoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced malignant disease (non-small cell lung cancer or malignant melanoma) (Experimental): Group 1: Participants with non-small cell lung cancer (NSCLC) as per inclusion/exclusion criteria undergo baseline PD-L1 expression testing by immunohistochemistry and [99m-Tc]-anti-PD-L1 single-domain antibody SPECT/CT imaging at 0 and 9 weeks.
  FDG-PET/CT is also performed at baseline (0) and first follow-up (9) weeks scans, in addition to standard CT clinical imaging at 0, 9 and 18 weeks.
  Group 2: Participants with malignant melanoma (MM) as per inclusion/exclusion criteria undergo baseline PD-L1 expression testing by immunohistochemistry and [99m-Tc]-anti-PD-L1 single-domain antibody SPECT/CT imaging at 0 and 12 weeks.
  FDG-PET/CT is also performed as standard clinical imaging at baseline (0), first follow-up (12) weeks and 24 weeks.
  Interventions: Diagnostic Test: [99mTc]-NM-01 SPECT/CT

INTERVENTIONS:
Diagnostic Test: [99mTc]-NM-01 SPECT/CT — Technetium labelled anti-PD-L1 single-domain antibody (NM-01) single-photon emission computed tomography (SPECT)/CT

SUMMARY:
Measurement of PD-L1 expression in cancer to monitor treatment response.

A prospective non-blinded, single centre, single interventional arm diagnostic imaging study.

To determine the baseline level and variability within and between patients and tumour types of PD-L1 expression in melanoma and non-small cell lung cancer in immunotherapy naïve patients using [99mTc]-anti-PD-L1 SPECT/CT and immunohistochemistry.

DETAILED DESCRIPTION:
Using [99mTc]-labeled anti-PD-L1 single-domain antibody, this study aims to prospectively measure changes in PD-L1 expression determined with SPECT/CT imaging and correlate these changes with response to anti-PD(L)1 immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Patients with histologically confirmed NSCLC or melanoma scheduled for PD1/PDL1 immunotherapy alone or in combination with other systemic anti-cancer therapy.
* Willingness and ability to comply with scheduled study visits and tests.

Exclusion Criteria:

* Pregnant or lactating women
* Concomitant uncontrolled medical conditions
* Patients likely to require palliative radiotherapy within the first 12 weeks of treatment or radiotherapy to target lesion(s) received within preceding 42 days
* More than 3 months between IHC PDL1 and study recruitment
* Patients who have received other systemic anti-cancer therapy within preceding 14 days
* Prognosis less than 3 months
* Previous anticancer treatment with any checkpoint inhibitor or other immunotherapy, i.e. only immunotherapy naïve patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage change in PD-L1 expression (using [99mTc] SPECT) in NSCLC. | Up to 18 weeks
  PD-L1 expression reported by measurement of tumour:blood pool ratio and/or SUV of [99mTc]-anti-PD-L1-sdAb uptake on SPECT. Measurement at baseline and 9 weeks will be compared to determine % change.
  Standard clinical imaging assessment at 9 and 18 weeks used as comparators.
Percentage change in PD-L1 expression (using [99mTc] SPECT) in melanoma lesions. | Up to 24 weeks
  PD-L1 expression reported by measurement of tumour:blood pool ratio and/or SUV of [99mTc]-anti-PD-L1-sdAb uptake on SPECT. Measurement at baseline and 12 weeks will be compared to determine % change.
  Standard clinical imaging assessment at 12 and 24 weeks used as comparators.

SECONDARY OUTCOMES:
Report PD-L1 tumour expression (using [99mTc] SPECT) of immunotherapy naive participants compared to PD-L1 expression determine by standard immunohistochemistry. | Baseline
  Correlation between PD-L1 expression reported by measurement of tumour:blood pool ratio and/or SUV of [99mTc]-anti-PD-L1-sdAb uptake on SPECT and PD-L1 expression determined by standard of care immunohistochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Gary JR Cook, Principal Investigator — King's College London, London, UK
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hughes DJ, Chand G, Johnson J, Tegala R, Bailey D, Adamson K, Edmonds S, Meszaros LK, Moore AEB, Manickavasagar T, Ndagire S, Gennatas S, Georgiou A, Ghosh S, Josephs D, Karapanagiotou E, McLean E, Ting HH, Spicer J, Goh V, Cook GJR. PD-L1 imaging with [99mTc]NM-01 SPECT/CT is associated with metabolic response to pembrolizumab with/without chemotherapy in advanced lung cancer. Br J Cancer. 2025 Jun;132(10):913-921. doi: 10.1038/s41416-025-02991-w. Epub 2025 Apr 5. PMID 40188291
- [Derived] Hughes DJ, Chand G, Johnson J, Bailey D, Adamson K, Goh V, Cook GJR. Inter-rater and intra-rater agreement of [99mTc]-labelled NM-01, a single-domain programmed death-ligand 1 (PD-L1) antibody, using quantitative SPECT/CT in non-small cell lung cancer. EJNMMI Res. 2023 May 31;13(1):51. doi: 10.1186/s13550-023-01002-4. PMID 37256434
- [Derived] Nazir MS, Hughes DJ, Chand G, Adamson K, Johnson J, Bailey D, Gibson V, Ting HH, Lyon AR, Cook GJR; PECan study group. [99mTc]-labelled anti-Programmed Death-Ligand 1 single-domain antibody SPECT/CT: a novel imaging biomarker for myocardial PD-L1 expression. EJNMMI Res. 2023 May 17;13(1):44. doi: 10.1186/s13550-023-00990-7. PMID 37195370